CLINICAL TRIAL: NCT00510094
Title: Determining the Efficacy of a Relational Aggression Intervention for Urban African American Girls
Brief Title: Effectiveness of Treatment for Relational Aggression in Urban African American Girls
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-10-5013; R01MH075787 (NIH); DSIR 84-CTS
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Aggression
Keywords: Social Skills; Anger Management; Relational Aggression
MeSH Terms: conditions — Aggression; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive the Friend to Friend program
  Interventions: Behavioral: Friend to Friend program
- 2 (Active Comparator): Participants will receive the psychoeducational attention control intervention
  Interventions: Behavioral: Psychoeducational attention control intervention

INTERVENTIONS:
Behavioral: Friend to Friend program — Friend to Friend arm is a social information processing group treatment to help aggressive girls learn better social problem solving and decision making choices. Participants will learn how to identify signs of physiological arousal, evaluate others' intentions, react to a potential conflict situation, and generate and evaluate alternatives. Treatment sessions are twice per week (30 to 40 minutes per session) for ten weeks.
  Other Names: Relational aggression intervention
  Arms: 1
Behavioral: Psychoeducational attention control intervention — Psychoeducational attention control group also meets two times per week for 10 weeks to control for nonspecific factors of treatment. Participants learn homework, study skills, and organizational skills.
  Other Names: Homework and study skills intervention
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a school-based social cognitive group treatment in reducing aggression (bullying) among relationally aggressive urban African American girls.

DETAILED DESCRIPTION:
Relational aggression, also known as "female bullying," is a type of psychological aggression in which covert tactics are used to harm other people and their relationships. These tactics include humiliation, intimidation, coercing, shaming, malicious teasing, shunning, and using other forms of emotional abuse in an attempt to harm others. Although aggressive behavior is typically common among younger children, most children become less aggressive as they mature and develop better interpersonal skills. However, consistent aggressive behavior can lead to further problems and increased violence in the aggressor. In this study, a social cognitive anger management group intervention called Friend to Friend (F2F) will be evaluated as a way to develop more productive social and emotional functioning among relationally aggressive urban African American girls.

Participants will be randomly assigned to either the F2F program or a psycho-educational attention control (PAC) group. All participants will attend 40-minute treatment sessions twice a week for a total of 10 weeks. The sessions will occur during the girls' lunch or recess period. Participants assigned to the F2F program will learn how to identify signs of physiological arousal, react to a potential conflict while generating alternatives to the solution, and apply previously discussed social cognitive strategies to different situations. Culturally specific cartoons, videotape illustrations, and role playing will be used to portray these improved strategies and behaviors. Participants assigned to the PAC group will learn different organization and homework strategies as well as how to improve their study skills in an attempt to improve their overall academic performance. Outcomes will be assessed through observation, school reports, and questionnaires for all participants at baseline, immediately after treatment, and 9 months after treatment.

ELIGIBILITY:
Inclusion Criteria for Schools :

* Urban school located in Southwest Philadelphia
* Student body is more than 80% African American
* Large school with at least three classrooms per grade
* Not currently involved with systematic anti-aggression social skills program

Inclusion Criteria for Participants:

* In the 3rd, 4th, or 5th grade
* Meets diagnostic criteria for relational aggression

Exclusion Criteria for Participants:

* Enrolled in special education and not integrated into a regular education classroom

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-10; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Peer nominations | Measured pre-treatment and immediately post-treatment
Playground observations | Measured pre-treatment and immediately post-treatment
Children's Social Behavior Questionnaire | Measured pre-treatment and immediately post-treatment and at 9-month follow-up
Social Cognitive Assessment Profile | Measured pre-treatment and immediately post-treatment and at 9-month follow-up
Cartoon Based Hostile Attribution Bias Measure | Measured pre-treatment and immediately post-treatment and at 9-month follow-up
Knowledge of Anger Problem Solving (KAPS) | Measured pre-treatment, immediately post-treatment, and at 9 month follow-up

SECONDARY OUTCOMES:
Discipline referrals and suspensions | Measured pre-treatment, immediately post-treatment and at 9-month follow-up
Academic Performance Rating Scale | Measured pre-treatment, immediately post-treatment and at 9-month follow-up
Homework Performance Questionnaire | Measured pre-treatment, immediately post-treatment and at 9-month follow-up
Asher-Wheeler Loneliness Questionnaire | Measured pre-treatment, immediately post-treatment and at 9-month follow-up
Iowa-Conner Aggression subscale | Measured pre-treatment, immediately post-treatment and at 9-month follow-up
Student-Teacher Relationship Scale | Measured pre-treatment, immediately post-treatment and at 9-month follow-up
Peer Ratings of Aggression and Prosocial Behavior | Measured pre-treatment, immediately post-treatment
Harter, Self-Perception Profile for Children | Measured pre-treatment, immediately post-treatment, and at 9 month follow-up
Peer Sympathy Scale | Measured pre-treatment, immediately post-treatment, and at 9 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S. Leff, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Leff SS, Crick NR, Angelucci J, Haye K, Jawad AF, Grossman M, Power TJ. Social cognition in context: validating a cartoon-based attributional measure for urban girls. Child Dev. 2006 Sep-Oct;77(5):1351-8. doi: 10.1111/j.1467-8624.2006.00939.x. PMID 16999803
- [Background] Leff, S. S., Angelucci, J., Goldstein, A. B., Cardaciotto, L., Paskewich, B., & Grossman, M. (2007). Using a participatory action research model to create a school-based intervention program for relationally aggressive girls: The Friend to Friend Program. In J. Zins, M. Elias, & C. Maher (Eds.), Bullying, Victimization, and Peer Harassment: Handbook of Prevention and Intervention in Peer Harassment, Victimization, and Bullying (199-218). New York. Haworth Press.
- [Background] Leff SS, Gullan RL, Paskewich BS, Abdul-Kabir S, Jawad AF, Grossman M, Munro MA, Power TJ. An initial evaluation of a culturally adapted social problem-solving and relational aggression prevention program for urban African-American relationally aggressive girls. J Prev Interv Community. 2009;37(4):260-74. doi: 10.1080/10852350903196274. PMID 19830622
- [Background] Blom-Hoffman J, Leff SS, Franko DL, Weinstein E, Beakley K, Power TJ. Consent Procedures and Participation Rates in School-Based Intervention and Prevention Research: Using a Multi-Component, Partnership-Based Approach to Recruit Participants. School Ment Health. 2009 Mar 1;1(1):3-15. doi: 10.1007/s12310-008-9000-7. PMID 19834586
- [Background] Gullan RL, Feinberg BE, Freedman MA, Jawad A, Leff SS. Using Participatory Action Research to Design an Intervention Integrity System in the Urban Schools. School Ment Health. 2009 Sep 1;1(3):118-130. doi: 10.1007/s12310-009-9006-9. PMID 20428475
- [Background] Leff SS, Waasdorp TE. Effect of aggression and bullying on children and adolescents: implications for prevention and intervention. Curr Psychiatry Rep. 2013 Mar;15(3):343. doi: 10.1007/s11920-012-0343-2. PMID 23389773
- [Background] Waasdorp TE, Baker CN, Paskewich BS, Leff SS. The association between forms of aggression, leadership, and social status among urban youth. J Youth Adolesc. 2013 Feb;42(2):263-74. doi: 10.1007/s10964-012-9837-9. Epub 2012 Oct 20. PMID 23086015
- [Background] Macevoy JP, Leff SS. Children's sympathy for peers who are the targets of peer aggression. J Abnorm Child Psychol. 2012 Oct;40(7):1137-48. doi: 10.1007/s10802-012-9636-5. PMID 22556114
- [Background] Leff SS, Lefler EK, Khera GS, Paskewich B, Jawad AF. Preliminary examination of a cartoon-based hostile attributional bias measure for urban African American boys. Am J Community Psychol. 2012 Jun;49(3-4):332-46. doi: 10.1007/s10464-011-9461-y. PMID 21800228
- [Background] Leff SS, Waasdorp TE, Paskewich B, Gullan RL, Jawad AF, Macevoy JP, Feinberg BE, Power TJ. The Preventing Relational Aggression in Schools Everyday Program: A Preliminary Evaluation of Acceptability and Impact. School Psych Rev. 2010 Dec;39(4):569-587. PMID 21686034
- [Background] Leff SS, Cassano M, MacEvoy JP, Costigan T. Initial validation of a knowledge-based measure of social information processing and anger management. J Abnorm Child Psychol. 2010 Oct;38(7):1007-20. doi: 10.1007/s10802-010-9419-9. PMID 20449645